CLINICAL TRIAL: NCT04865809
Title: Professional and Home Oral Care With Non Surgical Periodontal Therapy for the Evaluation of Glycosylated Hemoglobin (HbA1c) in Patients Suffering From Diabetes Mellitus Type 1: a Randomized Clinical Trial.
Brief Title: Use of Ozonized Water With Toothpaste and Mousse in Non Surgical Periodontal Therapy for Patients With Diabetes Mellitus Type 1: a Randomized Clinical Trial.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pavia (Other)
Responsible Party: Principal Investigator, Andrea Scribante, Research Resident, Principal Investigator, University of Pavia
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2021-DIAB1
Record Dates: First submitted 2021-04-26; First posted 2021-04-29 (Actual); Last update posted 2022-03-29 (Actual); Status verified 2022-03

CONDITIONS: Diabetes Mellitus With Periodontal Disease
Keywords: ozonized water; glycosylated hemoglobin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Trial Group (Experimental): Patients from this group will use Peribioma Toothpaste and Mousse for home oral care.
  Interventions: Other: Peribioma Toothpaste and Mousse
- Control Group (Active Comparator): Patients from this group will use Biorepair Plus Parodontgel for home oral care.
  Interventions: Other: Standard toothpaste

INTERVENTIONS:
Other: Peribioma Toothpaste and Mousse — Use of Peribioma Toothpaste and Mousse for home oral care.
  Arms: Trial Group
Other: Standard toothpaste — Use of Biorepair Plus Parodontgel for home oral care
  Arms: Control Group

SUMMARY:
The aim of this study is to evaluate the efficacy of Peribioma Toothpaste and Mousse for home oral care in patients with Diabetes Mellitus Type 1.

Patients will undergo a professional oral hygiene procedure, followed by irrigation with ozonized water.

Patients will be randomly divided into two groups:

* Trial Group: patients will use Biorepair Peribioma Toothpaste and Mousse for home oral care
* Control Group: patients will use Biorepair Plus Parodontgel toothpaste for home oral care.

The variations of the following indices will be evaluated at the baseline, after 3 and 6 months: glycosylated hemoglobin (HbA1c) , Clinical Attachment Level (CAL), Plaque Index (PI), Probing Pocket Depth (PPD) and Bleeding on Probing (BoP).

DETAILED DESCRIPTION:
The aim of this study is to evaluate the efficacy of Peribioma Toothpaste and Mousse for home oral care in patients with Diabetes Mellitus Type 1.

Patients who respond to eligibility criteria and that will sign the informed consent will undergo a professional oral hygiene procedure; then, ozonized water (aquolab) will be used to irrigate periodontal pockets for 1 minute.

Then, patients will be randomly divided into two groups:

* Trial Group: patients will use Biorepair Peribioma Toothpaste and Mousse for home oral care until the end of the study;
* Control Group: patients will use Biorepair Plus Parodontgel toothpaste for home oral care until the end of the study.

Changes in the following indices will be evaluated at the baseline, after 3 and 6 months: glycosylated hemoglobin (HbA1c) , Clinical Attachment Level (CAL), Plaque Index (PI), Probing Pocket Depth (PPD) and Bleeding on Probing (BoP).

ELIGIBILITY:
Inclusion Criteria:

* patients suffering from Diabetes Mellitus Type 1
* adult patients
* patients who agreed to participate to the study and that signed the informed consent.

Exclusion Criteria:

* patients taking intravenous or oral Bisphosphonates at the study begin or in the previous 12 months
* patients with low compliance and motivation to participate
* pazienti irradiati alla testa o collo negli ultimi 12 mesi
* pregnant or breastfeeding women
* alcohol and drug abuse
* patients with psychiatric diseases

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2021-05-12 (Actual); Primary Completion 2022-01-13 (Actual); Study Completion 2022-01-16 (Actual)

PRIMARY OUTCOMES:
Change in Glycosylated Hemoglobin (HbA1c) | Baseline, 3 and 6 months.
  Serum levels of glycosylated hemoglobin
Change in CAL - Clinical Attachment Loss | Baseline, 3 and 6 months.
  Measurement (in mm) of the position of the gingival margin in relation to the cemento-enamel junction (CEJ).
Change in PI - Plaque Index (Silness and Löe, 1964) | Baseline, 3 and 6 months.
  Scoring criteria:
  0 = no plaque;
  1. = thin plaque layer at the gingival margin, only detectable by scraping with a probe;
  2. = moderate layer of plaque along the gingival margin; interdental spaces free, but plaque is visible to the naked eye;
  3. = abundant plaque along the gingival margin; interdental spaces filled with plaque.
Change in PPD - Probing Pocket Depth | Baseline, 3 and 6 months.
  Evaluation (in mm) of the depth of the gingival sulcus, through a millimeter periodontal probe; it is detected from the gingival margin to the bottom of the gingival sulcus or periodontal pocket, evaluated at 6 sites.
Change in BOP - Bleeding on Probing (percentage) | Baseline, 3 and 6 months.
  Site-specific assessment of the presence or absence of gum bleeding after the insertion of the periodontal probe for the detection of PPD, detected on 6 sites.
  Percentage of sites with bleeding on probing determines the BOP%.

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Scribante, DDS, PhD., Principal Investigator — University of Pavia
Locations (1):
- Unit of Dental Hygiene - Section of Dentistry - Department of Clinical, Surgical, Diagnostic and Paediatrics - University of Pavia, Pavia, Lombardy, Italy

IPD SHARING:
Plan to Share IPD: No
Data will be available upon motivated request to Principal Investigator